CLINICAL TRIAL: NCT04460651
Title: PREPARE-IT. Prevention and Treatment of COVID19 With EPA in Subjects at Risk - Intervention Trial
Acronym: PREPARE-IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Estudios Clínicos Latino América (Other)
Collaborators: Amarin Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PREPARE-IT. Version 4.0
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: COVID19
Keywords: Icosapent ethyl; Vascepa; Eicosapentaenoic acid ethyl ester; Ethyl-EPA; AMR101
MeSH Terms: conditions — COVID-19 | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Intervention Model Description: Simple, pragmatic, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active treatment (Active Comparator): Participants in this arm will receive study medication icosapent ethyl (IPE) with a specific dose scheme.
  Interventions: Drug: Icosapent ethyl (IPE)
- Placebo (Placebo Comparator): Participants in this arm will receive Placebo with the same dose scheme as the active comparator:
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Icosapent ethyl (IPE) — Participants in this arm will receive study medication IPE with the following dosage schedule:
  8 g of IPE (4 capsules every 12 hours - morning and evening, with food) for the first three days followed by 4 g of IPE (2 capsules every 12 hours - morning and evening, with food) thereafter (days 4-28 for treatment arm and 4-60 for prevention arm)
  Other Names: Vascepa®
  Arms: Active treatment
Drug: Placebo — Participants in this arm will receive placebo with the following dosage schedule: 8 g of placebo (4 capsules every 12 hours - morning and evening, with food) for the first three days followed by 4 g of placebo (2 capsules every 12 hours - morning and evening, with food) thereafter (days 4-28 for treatment arm and 4-60 for prevention arm)
  Arms: Placebo

SUMMARY:
The PREPARE-IT investigator-initiated trial program is a simple, pragmatic, therapeutic strategy evaluating pure icosapent ethyl (IPE) at initially higher doses intended to reduce infection rates and subsequent morbidity and mortality among subjects at high risk of infection due to COVID-19 (prevention arm), and to reduce the hospitalization rate and complications in patients with a positive diagnosis of COVID-19 (treatment arm).

DETAILED DESCRIPTION:
Few vaccines have received emergency authorization providing relative immunity, reducing both transmission and infection rates and subsequent associated morbidity and mortality. However, broad access to vaccines is limited globally, and emergence of COVID-19 viral mutations and vaccine breakthrough cases underscore the need for complementary effective therapies.

To date, there are limited systemic options available for effective treatment from viral-inhibitors, polyclonal antibodies (immunomodulatory drugs) to mitigate the inflammatory cascade and subsequent cytokine storm, and low-dose steroids such as dexamethasone in high-risk patients, which was associated with a reduction in mortality.

Icosapent ethyl (IPE) is a safe, well-tolerated oral therapy proven to be effective in improving outcomes in patients with established cardiovascular disease or diabetes with one or more additional risk factors.

In the context of COVID-19, a recent pilot study on 50 patients on a loading dose of 8g/day for three days, followed by 4g/daily showed a significant improvement in validated patient-reported FLU-PRO score symptoms. A corresponding reduction in a key biomarker of inflammation (hs-CRP) was also detected within the IPE arm at 14 days.

While this pilot study provides the first evidence of an early anti-inflammatory effect of IPE, to confirm these findings, we designed a randomized, placebo-controlled study program investigating IPE with a similar loading dose intended to reduce infection rates and subsequent morbidity and mortality among subjects at high risk of infection from SARS-CoV-2 (prevention arm), and to reduce the hospitalization rate and complications in patients with a positive diagnosis of COVID-19 (treatment arm).

ELIGIBILITY:
(A) Prevention arm:

Inclusion Criteria:

1. 18 years of age or older and
2. any subject that is circulating and exposed to the public

Exclusion Criteria:

1. Previously diagnosed with COVID-19
2. Positive pregnancy test at the time of study entry in potentially fertile women
3. Pregnant or breastfeeding women
4. Subject who has received one or more doses of any vaccine for Sars-Cov-2 or who is scheduled to be vaccinated within the next 60 days
5. Unable to provide informed consent
6. Clear contraindication to EPA
7. Known hypersensitivity to the study drug
8. Administration of a drug with anticoagulant effects (antiplatelet agents are allowed)
9. Hemorrhagic Diathesis

(B) Treatment arm:

Inclusion Criteria:

1. 40 years of age or older and
2. Covid 19 diagnosis confirmed with SARS Cov-2 test (RT-PCR) and
3. No more than 7 days from the onset of symptoms and
4. Without clear indication for hospitalization (1-2 in the WHO COVID-19 Descriptive Score).

Exclusion Criteria:

1. Hospitalized patient or with a clear indication of hospitalization for COVID-19
2. Pregnant or breastfeeding women
3. Lack of access to adequate means of communication via the web
4. Unable to provide informed consent
5. Clear contraindication to EPA
6. Known hypersensitivity to the study drug
7. Administration of a drug with anticoagulant effects (antiplatelet agents are allowed)
8. Hemorrhagic Diathesis

Subjects who fill out the pre-selection form will be evaluated and approved for admission to the clinical trial after confirming their entry criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4093 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
(A) Prevention Arm: SARS-CoV-2 positivity assesed up to day 60. | 60 days
  SARS-CoV-2 positive subjects are defined as subjects with positive tests for SARS-CoV-2 RT-PCR or for SARS-CoV-2 lgG antibodies after developing COVID-19 disease at any stage within the follow-up period (including those subjects with or without symptomatic COVID-19 evaluated before the final visit) or those individuals who test positive for SARS-CoV-2 RT-PCR or for SARS-CoV-2 lgG antibodies at the final visit (day 60).
(B) Treatment Arm: COVID 19 related hospitalization (indication for hospitalization per the blinded investigator or actual hospitalization) or death assessed up to 28 days | 28 days

SECONDARY OUTCOMES:
(A) Prevention Arm: High-sensitivity C-reactive Protein (mg/dL) change from baseline to day 60 (key secondary outcome) | baseline, 60 days
  Mean change from baseline will be computed
(A) Prevention Arm: Triglycerides (mg/dL) change from baseline to day 60 | baseline, 60 days
  Mean change from baseline will be computed
(A) Prevention Arm: FLU-PRO SCORE change from baseline to day 60 in a subset of subjects | baseline, 60 days
  Mean change from baseline will be computed
(B) Treatment Arm: COVID 19 related hospitalization or death assessed up to 28 days (key secondary outcome) | 28 days
(B) Treatment Arm: Alive and out of the hospital at 28 days. | 28 days
(B) Treatment Arm: In hospital length of stay assessed up to 28 days | 28 days
(B) Treatment Arm: New requirement of mechanical ventilation assed up to 28 days. | 28 days
(B) Treatment Arm: Total events: non-fatal myocardial infarction or non-fatal stroke or death (initial and subsequent), until day 28. | 28 days
(B) Treatment Arm: Total mortality assessed up to 28 days | 28 days
(B) Treatment Arm: FLU-PRO SCORE change from baseline at 28 days | (B) Treatment Arm:

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Diaz, MD, Principal Investigator — ECLA- Estudios Clínicos Latino América
Locations (1):
- Instituto de Investigaciones Clínicas - Rosario, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: No